CLINICAL TRIAL: NCT03874780
Title: First in Human (FIH) Study for the Evaluation of the Safety and Early Performance of the Vibe Delivery System for the Delivery of Botox™ in Subjects With Idiopathic Overactive Bladder (OAB)
Brief Title: Vibe First In Human Study for the Assessment of Safety and Initial Performance of the Vibe Delivery System in Subjects With Idiopathic Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vensica Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-100
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-03

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Subjects treated with Botox (TM) with the Vibe investigational delivery system
  Interventions: Device: Vibe Delivery system

INTERVENTIONS:
Device: Vibe Delivery system — delivery of Botox (TM) to the bladder wall using an ultrasound technology with the Vibe delivery system

SUMMARY:
This First In Human study is aimed to evaluate the safety and initial efficacy of the Vibe delivery system in delivering Botox (TM) to the bladder wall in patients diagnosed with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects between the ages of 18 to 80 years old diagnosed with idiopathic OAB.
2. Subject has signed Informed Consent Form and is willing and able to comply with all requirements of the protocol.
3. Subjects with symptoms of incontinence associated with OAB for ≥ 3 months prior to screening.
4. Subjects who are non-responsive, non-compliant or intolerable to pharmacologic oral therapy (e.g., anticholinergic agents).
5. Subject is willing and able to initiate self-catheterization post-treatment, if required.
6. Subjects with PVR ≤200 ml.
7. Subjects who are mentally competent, with the ability to understand and comply with the requirements of the study.
8. A negative urine pregnancy test during screening in women with childbearing potential. A female subject will also agree to use an adequate birth control method for the duration of her participation in the study and for a period of 6 months after participation completion.

Exclusion Criteria:

1. Subjects currently using Clean intermittent catheterization (CIC) or indwelling catheter to manage their urinary incontinence.
2. Pregnant or breastfeeding women, or women of childbearing potential who are planning to become pregnant during the study period or not practicing reliable contraception methods.
3. Subjects with clinically significant Bladder Outlet Obstruction (BOO) according to medical history.
4. Subjects with active urinary tract infection, as diagnosed on screening urinalysis.
5. Subjects with known polyuria or polydipsia.
6. Subjects with a known positive diagnosis of Myasthenia gravis, Eaton-Lambert syndrome, or Amyotrophic Lateral Sclerosis.
7. Subjects with OAB due to any known neurological reason.
8. Subjects currently undergoing biofeedback, pelvic muscle rehabilitation, pelvic floor physical therapy, or electrical-stimulation who are unwilling to discontinue such treatments for the duration of study participation.
9. Subject with a 24-hour total urine volume voided greater than 3,000 ml, as measured at screening visit.
10. Predominance of stress incontinence in the opinion of the investigator, determined by medical history.
11. Subjects with vesico-ureteral reflux, genitourinary fistulae.
12. Subjects with pelvic organ prolapse stage III or IV, (i.e. the most distal part of the prolapse protruding more than 1 cm beyond the hymen at straining).
13. Subjects with prior Botox™ therapy of any serotype within 12 weeks for any indication, including urologic condition.
14. Subjects with a history of pelvic radiation therapy.
15. Subject who is morbidly obese (BMI > 40 Kg/m2).
16. Subjects with a history of treatment for two or more UTIs within 6 months prior to screening or use of prophylactic antibiotics to prevent chronic UTIs.
17. Subjects on immunomodulatory therapy (suppressive or stimulatory).
18. History or evidence of any pelvic or lower tract genitourinary abnormalities, malignancy, bladder surgery (excluding stress incontinence or pelvic organ prolapse surgeries), or disease, other than OAB.
19. Subjects with operative sling erosion.
20. History of interstitial cystitis/painful bladder syndrome, in the opinion of the investigator.
21. Subjects with current major psychiatric disorder or other psychiatric or medical issues that would interfere with study participation (e.g. dementia, psychosis, upcoming major surgery, etc).
22. Subject has severe cardiac, pulmonary, renal, or hepatic disease that in the judgment of the study physician would preclude participation in this study.
23. Any other condition or medical history, that to the discretion of the investigator and/or Sponsor, excludes the subject from participation in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events Reporting | 7 days
  Incidence of device related SAEs

SECONDARY OUTCOMES:
Serious Adverse Events Reporting | 12 weeks
  Incidence of device related SAEs within
Incontinence | 12 weeks
  Change from Baseline in the mean number of Episodes of Urinary Incontinence/24h, as assessed by urinary diary
Micturition | 12 weeks
  Change from Baseline in frequency of Micturition Episodes/24h, as assessed by urinary diary
Nocturia | 12 weeks
  Change from Baseline in Daily Average Number of Nocturia Episodes, as assessed by urinary diary
Urgency | 12 weeks
  Change from baseline in Urinary urgency, as assessed by urinary diary

OTHER OUTCOMES:
Treatment Response | 12 weeks
  Percentage of subjects who have a Positive Treatment Response on the Treatment Benefit Scale (TBS)
Change in Quality of Life Total Score | 12 weeks
  Change from baseline in Overactive Bladder Quality of life (OAB-q) total score. The OAB-q questionnaire is a validated, multi-sectional questionnaire that assesses the patient's coping with overactive bladder symptoms. The questionnaire is commonly used in clinical research and clinical setting for this indication, and consists of the following 6 scores:
  * Symptoms severity score
  * Coping score
  * Concern/worry score
  * Social score
  * Sleep score
  * Quality of life score These scores are further analyzed to obtain two domains: Quality of Life total score (improvement is demonstrated in higher scores), and Symptoms Bother Score (improvement is demonstrated in lower scores).

CONTACTS AND LOCATIONS:
Overall Officials: ‪Maya Shick‬, Study Director — Consultant
Locations (2):
- Jablonec Nad Nisou Medical Center, Jablonec nad Nisou, Czechia
- Braga Medical Center, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No